CLINICAL TRIAL: NCT06709521
Title: Optimization of Beta-lactam Dosing in Critically Ill Patients With Suspected or Documented Antimicrobial Resistant Gram-Negative Infections With Cystatin-C (OPTIMIZE-GNI)
Brief Title: Optimization of Beta-lactam Dosing in Critically Ill Patients With Cystatin C (OPTIMIZE-GNI)
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-0013; 5UM1AI104681-12 (NIH)
Record Dates: First submitted 2024-10-31; First posted 2024-11-29 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-07-18

CONDITIONS: Bacterial Infection
Keywords: AMR; Beta-lactam; Cefepime; cystatin-C; eGFR; Gram-negative; Iohexol; Meropenem
MeSH Terms: conditions — Bacterial Infections | interventions — Iohexol

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Arm 1 (Experimental): Adult patients in the ICU receiving either meropenem or cefepime as part of their clinical management will receive one dose of IV iohexol 1500 mgI (5 mL) via slow push administration on Study Days 1 and 2 prior to the start of first or second daily meropenem or cefepime dose. N=150
  Interventions: Drug: Iohexol

INTERVENTIONS:
Drug: Iohexol — Iohexol,N,N´ -Bis(2,3-dihydroxypropyl)-5-[N-(2,3-dihydroxypropyl)-acetamido]-2,4,6-triiodoisophthalamide, is a non-ionic, water-soluble radiographic contrast medium with a molecular weight of 821.14 (iodine content 46.36%)

SUMMARY:
The purpose of this study is to evaluate the abilities of Cystatin C (CysC) and CysC-based estimated Glomerular Filtration Rate (eGFR) equations to characterize the pharmacokinetics (PK) profiles of meropenem and cefepime relative to Serum Creatinine (SCR), Serum Creatinine based Equation (SCRE)and iohexol at the population and individual levels in critically ill adult patients with suspected or documented AMR Gram-negative infections. We hypothesize that CysC and CysC-based eGFR equations will characterize the PK profiles of meropenem and cefepime at the population and individual levels with greater accuracy and precision than SCR and SCREs. Iohexol will be administered to patients enrolled in the study and serve as the reference indicator of measured Glomerular Filtration Rate (mGFR), which is the gold standard assessment of kidney function. We hypothesize that the predictive performances of CysC and CysC-based eGFR equations in estimating the PK profiles of meropenem and cefepime at the population and individual levels will be comparable to iohexol. The information obtained in this study will be used to develop PK/pharmacodynamics (PD) optimized meropenem and cefepime dosing schemes based on the renal function biomarker population PK (PopPK) model with the best predictive performance for clinical use in the treatment of critically ill adult patients with suspected or documented AMR Gram-negative infections and varying degrees of renal function. The primary objective of this study is to compare the abilities of renal function biomarkers (CysC, CysC-based eGFR equations, SCR, SCREs) relative to iohexol to characterize the PK profiles of meropenem and cefepime in critically ill adult patients with suspected or documented AMR Gram-negative infections.

DETAILED DESCRIPTION:
The intent of this study is to compare the abilities of Cystatin C (CysC) and CysC-based estimated Glomerular Filtration Rate (eGFR) equations to characterize the pharmacokinetics (PK) profiles of meropenem and cefepime relative to Serum Creatinine (SCR), Serum Creatinine based Equation (SCRE), and iohexol in critically ill patients with suspected or documented AMR Gram-negative infections. We hypothesize that CysC and CysC-based eGFR equations will characterize the PK profiles of meropenem and cefepime at the population and individual levels with greater accuracy and precision than SCR and SCREs. Iohexol will be administered to patients enrolled in the study and serve as the reference indicator of measured Glomerular Filtration Rate (mGFR), which is the gold standard assessment of kidney function. We further hypothesize that the predictive performances of CysC and CysC-based eGFR equations in estimating the PK profiles of meropenem and cefepime at the population and individual levels will be comparable to iohexol. Firstly, population PK (PopPK) modeling will be used to develop meropenem and cefepime PopPK models informed by CysC, CysC-based eGFR equations, SCR, and SCREs (renal function biomarkers), and iohexol. Secondly, model diagnostics will then be used to compare the predictive performances of the renal function biomarkers PopPK models for each antibiotic relative to iohexol PopPK model. Lastly, Monte Carlo simulation (MCS) will be used to design PK/ pharmacodynamics (PD) optimized meropenem and cefepime dosing schemes based on the renal function biomarker PopPK model with the best predictive performance for use in the treatment of critically ill adult patients with suspected or documented AMR Gram-negative infections and varying degrees of renal function. The primary objective of this study is to compare the abilities of renal function biomarkers (CysC, CysC-based eGFR equations, SCR, SCREs) relative to iohexol to characterize the PK profiles of meropenem and cefepime in critically ill adult patients with suspected or documented AMR Gram-negative infections. The secondary objective of this study is to develop PK/PD optimized meropenem and cefepime dosing schemes based on the renal biomarker function PopPK model with the best predictive performance relative to the iohexol PopPK model for critically ill adult patients with suspected or documented AMR Gram-negative infections.

ELIGIBILITY:
Inclusion Criteria:

1. Age >/=18 years at the time of enrollment.
2. Residing in an ICU.
3. Documented or suspected Antimicrobial Resistant (AMR) Gram-negative infection for which the prospective participant is receiving meropenem or cefepime as part of their clinical management.
4. Expectation that the prospective participant will reside in the ICU and receive meropenem or cefepime for the duration of the study, and that all study procedures will be completed.
5. Expectation that IV access will be sufficient for drug infusion and either IV or arterial access will be sufficient to allow for all protocol-required blood sampling to occur.
6. The prospective participant, or their legally authorized representative (LAR), is able and willing to provide signed informed consent

Exclusion Criteria:

1. Prospective participant has a documented hypersensitivity or allergic reaction to iohexol, any contrast agents, or iodine.
2. Prospective participant has a documented prior history of severe cutaneous reactions to iohexol, any contrast agents, or iodine.
3. Prospective participant received iohexol within one calendar day prior to enrollment or the expectation that they will receive iohexol for clinical care (i.e., Standard of Care [SOC]) during the study.
4. Prospective participant had a major surgery* within two calendar days prior to enrollment.

   *Major surgery will be defined as "the opening of either a body cavity or the mesenchymal barrier, using general anesthesia."
5. Prospective participant had a recent (within 6 months) burn involving > 25% of total body surface area.
6. Prospective participant had a penetrating injury* within two calendar days prior to enrollment.

   *Penetrating injury will be defined as an injury caused by a foreign object piercing the skin, which damages the underlying tissues and results in an open wound.
7. Prospective participant is currently receiving or is expected to receive any type of renal replacement therapy including hemodialysis or extra corporeal membrane oxygenation, during study period.
8. Prospective participant has a documented diagnosis of diabetes with a serum creatinine (SCR) obtained for clinical care purposes (i.e., SOC results) >3 mg/dL during screening.
9. Prospective participant has documented severe thyrotoxicosis as noted in medical records during screening.
10. Prospective participant is homozygous for sickle cell disease as noted in medical history/records.
11. Prospective participant has a documented diagnosis of hepatorenal syndrome as noted in medical records during screening.
12. Prospective participant is anuric* for >/ = 1 calendar day during screening AND has any one of the following documented conditions as noted in medical history/records:

    * Pheochromocytoma
    * Myelomatosis
    * Multiple myeloma
    * Paraproteinemia *Anuria is defined as urine production <100 mL in a calendar day
13. Prospective participant is pregnant or breastfeeding.
14. Prospective participant received or is expected to receive albumin from one calendar day prior to enrollment to end of study period.
15. Prospective participant received or is expected to receive >/= 3 units of any blood product other than platelets from one calendar day prior to enrollment to end of study period.
16. Any condition that, in the judgment of the investigator, precludes participation because it could affect the prospective participant's safety.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-02-12 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Akaike's information criterion (AIC) of cefepime | Days 1-2
  For PopPK models
Akaike's information criterion (AIC) of iohexol | Days 1-2
  For PopPK models
Akaike's information criterion (AIC) of meropenem | Days 1-2
  For PopPK models
Clearance (Cl) of cefepime | Days 1-2
Clearance (Cl) of iohexol | Days 1-2
Clearance (Cl) of meropenem | Days 1-2
Intercompartment rate constant of cefepime | Days 1-2
Intercompartment rate constant of iohexol | Days 1-2
Intercompartment rate constant of meropenem | Days 1-2
Objective function value (OFV) of cefepime | Days 1-2
  For PopPK models
Objective function value (OFV) of iohexol | Days 1-2
  For PopPK models
Objective function value (OFV) of meropenem | Days 1-2
  For PopPK models
Volume of distribution (Vd) of cefepime | Days 1-2
Volume of distribution (Vd) of iohexol | Days 1-2
Volume of distribution (Vd) of meropenem | Days 1-2

SECONDARY OUTCOMES:
Pharmacokinetic/pharmacodynamics (PK/PD) optimized meropenem and cefepime dosing schemes | Days 1-2
  For PopPK models

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Harbor UCLA Medical Center - Medicine - Infectious Diseases, Torrance, California
  - Torrance Memorial Medical Center, Torrance, California
  - Henry Ford Health System - Henry Ford Hospital, Detroit, Michigan
  - Corewell Health - Infectious Disease, Royal Oak, Michigan
  - Duke University Hospital - Infectious Diseases, Durham, North Carolina
  - East Carolina University - Infectious Diseases and Tropical/Travel Medicine Clinic, Greenville, North Carolina
  - University of Cincinnati College of Medicine - Division of Infectious Diseases, Cincinnati, Ohio
  - Oregon Health and Science University - Adult Infectious Diseases Clinic, Portland, Oregon
  - University of Pittsburgh - Medicine - Infectious Diseases, Pittsburgh, Pennsylvania
  - Carilion Roanoke Memorial Hospital, Roanoke, Virginia